CLINICAL TRIAL: NCT05032911
Title: Analysis of Sensorimotor Control in People With and Without Neck Pain Using Inertial Sensor Technology: Study Protocol for a Longitudinal Prospective Observational Study
Brief Title: Sensorimotor Control in People With and Without Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Other Study IDs: CEU-023
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Movement Disorders; Neck Pain
MeSH Terms: conditions — Movement Disorders; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic participants: Asymptomatic subjects should not present any pain in the cervical region during the last 3 months and no previous treatment for neck pain in order to be included in the study.
  Interventions: Diagnostic Test: sensorimotor control analysis using inertial sensor technology
- Neck pain patients: Patients with neck pain should have an intensity of pain of at least 3 points out of 10 on a Visual Analog Scale and a neck pain duration of at least 3 months of evolution. Neck pain could be from nonspecific mechanical origin, associated with whiplash or with a previous medical diagnosis of degenerative or inflammatory alterations of the cervical spine, associated or not with headache and pain in the shoulder region or the upper limb.
  Interventions: Diagnostic Test: sensorimotor control analysis using inertial sensor technology

INTERVENTIONS:
Diagnostic Test: sensorimotor control analysis using inertial sensor technology — Inertial Measurement Unit (IMU) sensors will measure sensorimotor control variables including active range of motion, movement speed, acceleration, smoothness of motion, head repositioning accuracy and motion coupling patterns

SUMMARY:
This is a descriptive, observational, longitudinal, prospective study consecutively enrolling patients with non-specific neck pain and age-matched asymptomatic participants.

The investigators will register sensorimotor control variables, including active range of motion, movement speed, acceleration, smoothness of motion, head repositioning accuracy and motion coupling patterns. These variables will be recorded by means of Inertial Measurement Unit (IMU) sensors during the following tests consecutively performed in two measuring sessions separated by 12 months: (a) kinematics of planar movements, (b) kinematics of the craniocervical flexion movement, (c) kinematics during functional tasks and (d) kinematics of task-oriented neck movements in response to visual targets.

ELIGIBILITY:
Inclusion Criteria:

* Population aged between 18 and 65 years old

Exclusion Criteria:

* Visual impairment not corrected by the use of glasses/contact lenses
* Migraine headache
* Complex regional syndrome
* Previous surgeries in the neck and/or head region
* Sensory and/or vestibular alterations, (f) Otogenic or idiopathic vertigo/dizziness
* Presence of tumors in the craniocervical region
* Previous fracture in the head or neck region
* Osseous deformities in the thoracic, cervical or cranial region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from a community sample in Madrid, Spain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Active range of motion | 1 year
  Expressed as an angular displacement (°) in 3 full-movements (flexion-extension, lateral flexion and rotation)
Movement speed | 1 year
  Expressed as angular velocity (°/sec) in 3 full-movements (flexion-extension, lateral flexion and rotation)
Smoothness of motion | 1 year
  expressed as movement jerk (º/sec3)
Head repositioning accuracy | 1 year
  Calculated as the repositioning error considering the difference between the neutral starting position and the following positions reached after the performance of any of the movements
Motion coupling patterns | 1 year
  Calculated as the angular displacement occurring in a different anatomical plane to the one that is being tested for each of the planar movements

SECONDARY OUTCOMES:
Physical activity level | 1 year
  Measured using the short version of the International Physical Activity Questionnaire (IPAQ). The score of the scale is expressed in MET level x minutes of activity/day x days per week. Levels of 3.3 METs are considered light, 4.0 METs are moderate and 8.0 METs are vigorous.
Fear of movement and injury | 1 year
  Measured using the Tampa Scale for Kinesiophobia (TSK-11). It consists of 11 questions scored from 1 to 4. Therefore, a score of 11 is the lowest possible level of kinesiphobia, while 44 is the highest.
Pain-related fear-avoidance | 1 year
  Measured using the Fear Avoidance Components Scale (FACS). It has 20 itemsmeasured on a 6-point Likert scale for total possible score of 100 and the lowest possible score of 0. Higher scores indicate higher levels of fear avoidance.

REFERENCES:
- [Derived] Moggioli F, Perez-Fernandez T, Liebana S, Corredor EB, Armijo-Olivo S, Fernandez-Carnero J, Raya R, Conde P, Rodriguez-Lopez O, Sanchez C, Martin-Pintado-Zugasti A. Analysis of sensorimotor control in people with and without neck pain using inertial sensor technology: study protocol for a 1-year longitudinal prospective observational study. BMJ Open. 2022 Feb 15;12(2):e058190. doi: 10.1136/bmjopen-2021-058190. PMID 35168985